CLINICAL TRIAL: NCT00853970
Title: Efficacy Study of Bromfenac Ophthalmic Solution in Patients Undergoing Cataract Surgery
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bausch & Lomb Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CL-S&E-1205081-P
Record Dates: First submitted 2009-02-26; First posted 2009-03-02 (Estimated); Results first posted 2011-01-26 (Estimated); Last update posted 2013-01-25 (Estimated); Status verified 2013-01

CONDITIONS: Pain; Inflammation
Keywords: Pain and Inflammation as a function of cataract surgery
MeSH Terms: conditions — Pain; Inflammation

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Bromfenac ophthalmic solution 0.09% (Experimental): dosed 1 drop daily in study eye for 2 weeks
  Interventions: Drug: Bromfenac Ophthalmic Solution
- Placebo (Placebo Comparator): dosed 1 drop daily in study eye for 2 weeks
  Interventions: Drug: Placebo Comparator

INTERVENTIONS:
Drug: Bromfenac Ophthalmic Solution — sterile ophthalmic solution
  Arms: Bromfenac ophthalmic solution 0.09%
Drug: Placebo Comparator — sterile ophthalmic solution
  Arms: Placebo

SUMMARY:
Efficacy study of Bromfenac Ophthalmic Solution in cataract surgery

ELIGIBILITY:
Inclusion Criteria:

* Male or female at least 18 years of age who are scheduled for unilateral cataract surgery

Exclusion Criteria:

* Have known hypersensitivity to bromfenac or to any component of the investigational product

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 299 (Actual)
Dates: Start 2009-02; Primary Completion 2009-09 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tim McNamara, PharmD, Study Director — ISTA Pharmaceuticals, Inc.
Locations (1):
- ISTA Pharmaceuticals, Inc., Irvine, California, United States

REFERENCES:
- [Derived] Silverstein SM, Cable MG, Sadri E, Peace JH, Fong R, Chandler SP, Gow JA, Klier SM, McNamara TR; Bromfenac Ophthalmic Solution Once Daily (Bromday) Study Group. Once daily dosing of bromfenac ophthalmic solution 0.09% for postoperative ocular inflammation and pain. Curr Med Res Opin. 2011 Sep;27(9):1693-703. doi: 10.1185/03007995.2011.597663. Epub 2011 Jul 14. PMID 21751945

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The first participant entered the study on 02/09/2009, and last participant exited the study on 07/06/2009. This study took place at 41 sites in the USA
Pre-assignment Details: 152 participants were randomized to the bromfenac ophthalmic solution 0.09% treatment group and 147 were randomized to the placebo treatment group. One hundred forty six of 152 participants (96.1%) in the bromfenac ophthalmic solution 0.09% treatment group and 144/147 (98.0%) participants in the placebo treatment group completed the study.
Groups:
- Bromfenac Ophthalmic Solution 0.09%; Placebo: dosed 1 drop daily into the study eye for 2 weeks
Period: Overall Study
Arm/Group | Bromfenac Ophthalmic Solution 0.09% | Placebo
Started | 152 | 147
Completed | 146 | 144
Not Completed | 6 | 3
Not completed — Withdrawal by Subject | 2 | 1
Not completed — Cancelled surgery | 4 | 2

BASELINE CHARACTERISTICS:
Groups:
- Bromfenac Ophthalmic Solution 0.09%; Placebo: one drop daily in study eye for 2 weeks
- Total: Total of all reporting groups
Arm/Group | Bromfenac Ophthalmic Solution 0.09% | Placebo | Total
Number analyzed (Participants) | 152 | 147 | 299
Age Continuous [Mean (Full Range); unit: years] | 70.4 [34.0 to 87.0] | 69.1 [40.0 to 90.0] | 69.8 [34.0 to 90.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 89 | 99 | 188
  Male | 63 | 48 | 111

OUTCOME MEASURES:

1. Primary Outcome: Summed Ocular Inflammation Score (SOIS) of Zero
Description: Participants with SOIS of 0. Measured on a scale of 0-4: 0=0 cells (complete absence); 0.5=1-5 cells ; 1=6-15 cells (very slight); 2=16-25 cells (moderate); 3=26-50 cells (marked); 4=>50 cells (intense)
Time Frame: Day 15 (Primary Endpoint)
Population: Last observation carried forward (LOCF) Analysis; Intent to treat (ITT) Population
Measure: Number; unit: participants
Arm/Group | Bromfenac Ophthalmic Solution 0.09% | Placebo
Number analyzed (Participants) | 152 | 147
participants | 70 | 36

2. Secondary Outcome: Pain Free
Description: Participants that are pain free at day 1, taken from patient questionnaire with multiple possible responses measured on a scale of 0-3, where 0=none and 3=severe.
Time Frame: Day 1
Population: Last observation carried forward (LOCF) Analysis, Intent to treat (ITT) Population
Measure: Number; unit: participants
Arm/Group | Bromfenac Ophthalmic Solution 0.09% | Placebo
Number analyzed (Participants) | 152 | 147
participants | 135 | 105

ADVERSE EVENTS:
Time Frame: 2 weeks
Arm/Group | Bromfenac Ophthalmic Solution 0.09% | Placebo
Serious Adverse Events (participants affected / at risk) | 0/147 | 3/144
Other Adverse Events (participants affected / at risk) | 69/147 | 86/144
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Bromfenac Ophthalmic Solution 0.09% (N=147) | Placebo (N=144)
Acute and chronic pancreatitis (Endocrine disorders) | 0/146 (0) | 1 (1)
Eye and ear procedural complications (Surgical and medical procedures) | 0/146 (0) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bromfenac Ophthalmic Solution 0.09% (N=147) | Placebo (N=144)
Conjunctival hyperemia (Eye disorders) | 7 (7) | 9 (10)
Lacrimation increased (Eye disorders) | 5 (5) | 11 (11)
Eye Pain (Eye disorders) | 13 (15) | 34 (37)
Eye Inflammation (Eye disorders) | 15 (15) | 21 (22)
Foreign body sensation (Eye disorders) | 18 (21) | 20 (20)
Blurred Vision (Eye disorders) | 15 (15) | 11 (11)
Ocular Hyperemia (Eye disorders) | 4 (4) | 15 (18)
Photophobia (Eye disorders) | 11 (11) | 26 (26)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The disclosure restriction on the PI is that the PI will provide to the sponsor a copy of proposed publication information for review, comment and approval following completion of the study and at least sixty (60) days prior to submission of the publication. If sponsor requests in writing, the PI will withhold publication until written permission is given by Sponsor.